CLINICAL TRIAL: NCT04841213
Title: Prosthetics Dental Implant-based Rehabilitation in Patients With Loss of Teeth and Mineral Metabolism Disorders Due to Vitamin D3 Imbalance
Brief Title: Dental Implants Rehabilitation in Patients With Vitamin D3 Imbalance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13081986
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Tooth Loss; Vitamin D3 Deficiency; Osteomalacia
Keywords: tooth loss; vitamin D3 deficiency; dental implantation
MeSH Terms: conditions — Tooth Loss; Osteomalacia | interventions — Dental Implantation

STUDY DESIGN:
Intervention Model Description: Interventional retrospective prospective randomized clinical trial (RCT) in parallel groups.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Surgeons will be blinded to the endocrinologic status of patients who underwent or will undergo the dental implantation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group after vitamin D3 level stabilization (Active Comparator): Patients with loss of teeth and mineral metabolism disorders due to vitamin D3 imbalance (n=192) who will undergo dental implant placement after stabilization of vitamin D3 levels
  Interventions: Procedure: Dental implantation
- Group before vitamin D3 level stabilization (Active Comparator): Patients with the loss of teeth and mineral metabolism disorders due to vitamin D3 imbalance (n=192) who undergo the dental implantation during treatment by an endocrinologist
  Interventions: Procedure: Dental implantation

INTERVENTIONS:
Procedure: Dental implantation — Traditional 2-stage dental implantation according to surgical protocols of dental implant systems (Straumann (Institut Straumann AG, Switzerland), Astra Tech (Dentsply Implant Manufacturing GmbH, Germany), Xive (FRIADENT GmbH, Germany), Alpha Bio (Alpha Bio Tec Ltd., Israel) for different types of bone tissue
  Other Names: Bone plasty

SUMMARY:
Interventional retrospective prospective randomized clinical trial (RCT) in parallel groups.

The sample size is 384 patients with loss of teeth and vitamin D imbalance. All patients will undergo or underwent dental implantation after additional investigations which reveal vitamin D imbalance (<30 ng/ml or <75 nmol/l).

The 1 group will include 192 patients who will be or were operated on with dental implants after stabilization of vitamin D level with a help of an endocrinologist.

The 2 group will include 192 patients who will be or were operated on during the treatment of vitamin D imbalance prescribed by the endocrinologist.

The possible difference between groups can be considered the change of dental implants survival time and bone resorption level depending on the level of vitamin D and treatment time by the endocrinologist.

DETAILED DESCRIPTION:
A purpose is to increase the efficiency of rehabilitation of patients with loss of teeth and mineral metabolism disorders due to vitamin D3 imbalance using an interdisciplinary approach to dental implantation.

Retrospective prospective RCT in parallel groups includes 384 patients with loss of teeth and vitamin D3 imbalance who will undergo or underwent the dental implantation on the base of Oral Surgery Department of Borovskiy Institute of Dentistry of I.M.Sechenov First Moscow State Medical University (Sechenov University) and private dental clinic 'Society with limited responsibility (SLR) Topaz 2000' from 2010 till the 2021 year: prospective part will include 100 patients, the retrospective part will include 284 patients.

The counted sample size according to loss of teeth prevalence in Russia on the base of Sechenov University and private dental clinic Topaz 2000 is equal to 384 patients.

Randomization will be assured by surgeons blinded to endocrinologic status of patients who underwent or will undergo the dental implantation.

All patients will be included in 2 groups: 1 group will include patients (n=192), 25-50-years-old, with loss of teeth and mineral metabolism disorders due to vitamin D3 imbalance (<30 ng/ml, or <75 nmol/l) who will undergo dental implant placement after stabilization of vitamin D3 levels (>30-60 ng/ml, or 75-150 nmol/l for the process of treatment and monitoring); 2 group will include patients, 25-50-years-old, with the loss of teeth and mineral metabolism disorders due to vitamin D3 imbalance (n=192) who will undergo the dental implantation during treatment by an endocrinologist before the stabilization of vitamin D3 level in the blood.

Group 1

Patients will be directed for lab tests to detect mineral imbalance (vitamin D, ng/ml; parathyroid hormone (PH), thyroperoxidase antibodies (anti-TPO), Thyrotoxin 3 free (TT), Thyrotropic hormone (TH) pg/l) before dental implantation, and according to results, we will discuss further plan treatment with the endocrinologist. If it is needed due to the indications (adults with osteoporotic fractures; adults with a disease or condition accompanied by reduced bone mass or bone loss; all persons in the appointment of drug therapy, iatrogenic in relation to loss of bone mass; all patients receiving anti-osteopathic treatment to monitor its effectiveness; all persons who are not yet receiving treatment, but who may need it in case of bone loss.), Dual-Energy X-Ray Absorptiometry (DEXA) of skeleton mineral bone density will be done. After appropriate systemic treatment with vitamin D3 in 2 months after stabilization (>30 ng/ml, or >75 nmol/l) ) of vitamin D3 level (Aquadetrim (cholecalciferol) 15000 International Units (IU), Medana Pharma S.A., Poland, Registration number P N014088/01 from 21st June 2017; first 2 months taking orally 2-5 drops with a spoon of water depending on the severity of diseases, after 2 months and reaching the reference level of vitamin D its dose will be 1 drop per a day whole period of monitoring) the dental implantation was and will be performed with the further control of bone density and peri-implant tissues in 3 months after the operation. In the case of low bone density (type 3 or 4) the additional bone plasty was and will be performed. we assess the stability of dental implant on the stages of prosthetic rehabilitation according to the force of osteointegration during the inserting of the healing abutment (in Newtons on square centimeter), and each 1 year after treatment in the condition of periodical monitoring of patients with the endocrinologist (after the beginning of treatment after 2 months, then 1 time per 6 months).

Traditional 2-stage dental implantation will be performed according to surgical protocols of dental implant systems (Straumann (Institut Straumann AG, Switzerland, registration in Russia 03/10/2017 No FSZ 2010/06855), Astra Tech (Dentsply Implant Manufacturing GmbH, Germany, registration in Russia 27/09/2018 No FSZ 2008/02570), Xive (FRIADENT GmbH, Germany, registration in Russia 09/09/2008 No FSZ 2008/02568), Alpha Bio (Alpha Bio Tec Ltd., Israel, registration in Russia 26/04/2017 No FSZ 2009/05582), for different types of bone tissue

Group 2

Patients will be directed for lab tests to detect mineral imbalance (vitamin D, ng/ml; PH, anti-TPO, TT, TH, pg / l) before dental implantation, and according to results, we will discuss further plan treatment with the endocrinologist. If it is needed due to the indications (adults with osteoporotic fractures; adults with a disease or condition accompanied by reduced bone mass or bone loss; all persons in the appointment of drug therapy, iatrogenic in relation to loss of bone mass; all patients receiving anti-osteopathic treatment to monitor its effectiveness; all persons who are not yet receiving treatment, but who may need it in case of bone loss.), Dual-Energy X-Ray Absorptiometry (DEXA) of skeleton mineral bone density will be done. Treatment with vitamin D3 for stabilization of its level (>30 ng/ml, or >75 nmol/l) will be provided with Aquadetrim (cholecalciferol) 15000 International Units (IU), Medana Pharma S.A., Poland, Registration number P N014088/01 from 21st June 2017; first 2 months taking orally 2-5 drops with a spoon of water depending on the severity of diseases, after 2 months and reaching the reference level of vitamin D its dose will be 1 drop per a day whole period of monitoring). The dental implantation was and will be performed with the further control of bone density and peri-implant tissues in 3 months after operation at the beginning of treatment by endocrinologist without waiting of reference level of vitamin D. In case of low bone density of jaws (type 3 or 4) the additional bone plasty was or will be performed. We will assess the stability of dental implant on the stages of prosthetic rehabilitation according to the force of osteointegration during the inserting of the healing abutment (in Newtons on square centimeter), and each 1 year after treatment in the condition of periodical monitoring of patients with the endocrinologist (after the beginning of treatment after 2 months, then 1 time per 6 months)

Traditional 2-stage dental implantation according to surgical protocols of dental implant systems (Straumann (Institut Straumann AG, Switzerland, registration in Russia 03/10/2017 No FSZ 2010/06855), Astra Tech (Dentsply Implant Manufacturing GmbH, Germany, registration in Russia 27/09/2018 No FSZ 2008/02570), Xive (FRIADENT GmbH, Germany, registration in Russia 09/09/2008 No FSZ 2008/02568), Alpha Bio (Alpha Bio Tec Ltd., Israel, registration in Russia 26/04/2017 No FSZ 2009/05582), will be performed for different types of bone tissue

ELIGIBILITY:
Inclusion Criteria:

1. Signing of written informed consent of the patient to participate in a study
2. Age from 25 to 50 years old
3. Established diagnosis: tooth loss (K08.1- ICD 10), vitamin D3 imbalance.
4. Patients who are medically stable

Exclusion Criteria:

1. Refusal of the patient from further participation in the study
2. Pregnancy diagnosed after the inclusion into the trial
3. Non-compliance by the patient with postoperative recommendations.
4. Residence address change

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Primary Stability of dental implant | Day 0
  It can be assessed with the volume of torque during dental implant insertion with the physio-dispenser according to its program
Secondary Stability of dental implants after surgery | Days 60-90
  During the inserting of healing abutment the stability of dental implant will and was measured with the help of device Penguin RFA (Integration Diagnostics, Sweden, Registration 29th of December 2017 RZN No 2017/6664) (Quotient of stability depends on the scale from 1 to 99 ) based on resonance frequency analysis through the handpiece of device MulTipeg. The use of device will not and did not lead to the loss or mobility of dental implants.

SECONDARY OUTCOMES:
Colour of peri-implant tissues according to clinical examination after surgery | Days 3-7
  The condition of peri-implant tissues will be assessed according to their colour (points 0-1, where 0 - normal colour, 1- redness).
Oedema of peri-implant tissues according to clinical examination after surgery | Days 3-7
  The condition of peri-implant tissues will be assessed according to oedema volume (points 0-2, where 0- absence of oedema, 1- average oedema, 2 -intensive oedema in comparison to adjunct tissues condition)
Colour of peri-implant tissues according to clinical examination after surgery (for additional operations such bone plasty) | Days 10-14
  The condition of peri-implant tissues will be assessed according to their colour (points 0-1, where 0 - normal colour, 1- redness).
Oedema of peri-implant tissues according to clinical examination after surgery (for additional operations such bone plasty) | Days 10-14
  The condition of peri-implant tissues will be assessed according to oedema volume (points 0-2, where 0- absence of oedema, 1- average oedema, 2 -intensive oedema in comparison to adjunct tissues condition)
Colour of peri-implant tissues | Days 365-366
  The condition of peri-implant tissues will be assessed according to their colour (points 0-1, where 0 - normal colour, 1- redness).
Peri-implant pockets presence according to clinical examination | Days 365-366
  The condition of peri-implant tissues will be assessed according to presence of peri-implant pockets during probing (mm).
Condition of peri-implant tissues according to X-ray or cone-bean computed tomography | Days 365-366
  The condition of peri-implant tissues will be assessed according to presence of peri-implant pockets during radiological investigation (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Diachkova, PhD, Principal Investigator — I.M.Sechenov First Moscow State Medical University (Sechenov University)
Locations (2):
- Russia (2):
  - prof. Tarasenko Svetlana, Moscow
  - Vladimir Grachev, Moscow

IPD SHARING:
Plan to Share IPD: No
No, according to the rules (SOPs) of the Local Ethics Committee

REFERENCES:
- [Result] Diachkova E, Abramova EV, Blagushina NA, Tarasenko S. Surgical treatment with dental implants in a patient with secondary loss of teeth and osteoporosis caused by an imbalance of vitamin D. BMJ Case Rep. 2020 Nov 30;13(11):e235585. doi: 10.1136/bcr-2020-235585. PMID 33257353